CLINICAL TRIAL: NCT00584298
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Crossover Study in Women With Irritable Bowel Syndrome to Evaluate Feasibility and Reproducibility of Barostat Assessments of Colorectal Sensation During Colorectal Distention and Its Pharmacological Modulation Using Octreotide.
Brief Title: Feasibility and Reproducibility of Barostat Assessments of Colorectal Sensation During Colorectal Distention and Its Pharmacological Modulation Using Octreotide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CSMS995A2101
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Barostat; distention; IBS; irritable; bowel; syndrome; colorectal; sensation; modulation; reproducibility
MeSH Terms: conditions — Irritable Bowel Syndrome; Dilatation, Pathologic; Syndrome | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SMS995
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SMS995
  Other Names: Octreotide, Sandostatin
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study is designed to provide information on feasibility and reproducibility of barostat assessments of colorectal sensory functions and compliance and their pharmacological modulation

ELIGIBILITY:
Inclusion Criteria:

* A positive diagnosis of IBS.
* Subjects must either have been surgically sterilized, hysterectomized at least 6 months prior to screening, be postmenopausal or be using a double-barrier local
* contraception.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent

Exclusion Criteria:

* History of or evidence for structural diseases/conditions that affect the gastrointestinal system.
* Other diseases or conditions that in the opinion of the Investigator significantly affect colorectal sensitivity.
* Evidence of occult blood at stool analysis, or history of rectal bleeding.
* Using or planning to use drugs or agents during the study period that alter GI physiology and visceral perception.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
- 5 sensory pressure thresholds [mmHg] from ascending method of limits (AML) barostat protocol. - 16 sensory intensity ratings from the random phasic distention (RPD) barostat protocol. | throughout the study

SECONDARY OUTCOMES:
- colorectal compliance | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (7):
- United States (2):
  - Novartis Investigator Site, Boston, Massachusetts
  - Novartis Investigator Site, Rochester, Minnesota
- Novartis Investigator Site, Hamilton, Canada
- Novartis Investigator Site, Gothenburg, Sweden
- United Kingdom (3):
  - Novartis Investigator Site, London
  - Novartis Investigator Site, Manchester
  - Novartis Investigator Site, Nottingham